CLINICAL TRIAL: NCT01061164
Title: A Prospective Surveillance Study of Long-Term Outcomes in HIV-Infected Infants, Children and Adolescents
Brief Title: IMPAACT P1074: Long-Term Outcomes in HIV-Infected Infants, Children, and Adolescents
Status: Completed | Type: Observational
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: IMPAACT P1074; U01AI068632 (NIH)
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2014-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HIV-infected infants, children, and adolescents: Infants, children, and adolescents with HIV infection who have participated in PACTG 219C and/or select IMPAACT studies.

SUMMARY:
This study will examine the long-term effects of HIV infection, highly active antiretroviral therapy (HAART), and experimental treatments on children who participated in PACTG 219C or select IMPAACT studies.

DETAILED DESCRIPTION:
The use of HAART has been important in extending the lives of people with HIV infection. However, prolonged use of HAART may have long-term consequences. In addition, people participating in clinical trials using experimental therapies to treat HIV infection may experience negative health outcomes. The purpose of this study is to identify the long-term effects of HIV infection, HAART, and experimental treatments in infants, children, and adolescents.

This study will enroll children who participated in PACTG 219C or various IMPAACT studies. There will be no study visits specifically for this study. Researchers will review participants' medical records annually and collect information on illnesses, medications, CD4 cell count and viral load data, and body measurements.

ELIGIBILITY:
Inclusion Criteria:

* Past or current documentation of a confirmed diagnosis of HIV-1 infection defined as two separate peripheral blood specimens from different days, and each specimen must be positive. More information on this criterion can be found in the protocol.
* HIV-infected infants, children, or adolescents who participated in PACTG 219C during 5/1/06-5/31/07 and are not currently participating in ongoing long-term follow-up (LTFU) studies (e.g., Pediatric HIV/AIDS Cohort Study Adolescent Master Protocol [PHACS AMP], LEGACY). Please refer to the IMPAACT website for the current list of studies or contact the protocol team (actg.teamp1074@fstrf.org).

OR

* HIV-infected infants, children, and adolescents at domestic sites who have participated in or are currently participating in IMPAACT treatment studies (including studies that have rolled over from the PACTG into IMPAACT) designated by the IMPAACT Network Executive Committee (NEC) for subsequent LTFU in this study, and are not currently participating in ongoing LTFU studies. Please refer to the IMPAACT website for the current list of studies or contact the protocol team (actg.teamp1074@fstrf.org).
* Parent or legally-accepted representative/guardian is able and willing to provide signed informed consent for minors (unless child has emancipated minor status)

Exclusion Criteria:

* Current participation in other ongoing LTFU studies (e.g., PHACS AMP, LEGACY). Please refer to the IMPAACT website for the current list of studies or contact the protocol team (actg.teamp1074@fstrf.org).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include participants in PACTG 219C or select IMPAACT treatment studies.
Sampling Method: Non-Probability Sample
Enrollment: 1207 (Actual)
Dates: Start 2009-03; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To identify possible long-term adverse outcomes of HIV infection and complications of antiretroviral therapy (ART) or experimental interventions other than ARTs in HIV-infected infants, children, and adolescents at IMPAACT sites in the United States | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Myron J. Levin, MD, Study Chair — University of Colorado at Denver Health Sciences Center; Paige L. Williams, PhD, Study Chair — Harvard School of Public Health (HSPH)
Locations (39):
- United States (37):
  - Univ. of Alabama Birmingham NICHD CRS (5096), Birmingham, Alabama
  - Miller Children's Hospital Long Beach (5093), Long Beach, California
  - Usc La Nichd Crs (5048), Los Angeles, California
  - Childrens Hospital Los Angeles (5090), Los Angeles, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CR (3601), Los Angeles, California
  - UCSD Mother, Child & Adolescent HIV Program(4601), San Diego, California
  - Univ. of California San Francisco NICHD CRS (5091), San Francisco, California
  - University of Colorado Denver NICHD CRS (5052), Aurora, Colorado
  - Children's National Med. Ctr. Washington DC NICHD CRS (5015), Washington D.C., District of Columbia
  - Howard University Washington DC NICHD CRS (5044), Washington D.C., District of Columbia
  - South Florida CDC Ft Lauderdale NICHD CRS (5055), Fort Lauderdale, Florida
  - Univ. of Florida Jacksonville NICHD CRS (5051), Jacksonville, Florida
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS (4201), Miami, Florida
  - University of South Florida Tampa (5018), Tampa, Florida
  - Chicago Children's CRS (4001), Chicago, Illinois
  - Tulane University (5095), New Orleans, Louisiana
  - Johns Hopkins University NICHD CRS (5092), Baltimore, Maryland
  - Children's Hospital of Boston NICHD CRS (5009), Boston, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS (7301), Worcester, Massachusetts
  - Wayne State University/Children's Hospital of Michigan NICHD CRS (5041), Detroit, Michigan
  - New Jersey Medical School (NJ) (2802), Newark, New Jersey
  - Univ of Med & Dentistry of New Jersey/Univ Hosp, Newark, New Jersey
  - New York University NY (5012), New York, New York
  - Metropolitan Hospital (5003), New York, New York
  - Columbia IMPAACT Center (4101), New York, New York
  - Strong Memorial Hospital, University of Rochester NICHD CRS (5057), Rochester, New York
  - SUNY Stony Brook (5040), Stony Brook, New York
  - Bronx-Lebanon Hospital IMPAACT CRS (6901), The Bronx, New York
  - Jacobi Medical Center Bronx (5013), The Bronx, New York
  - Duke Pediatric Infectious Diseases, Durham, North Carolina
  - Duke University Medical Center (DUMC) Pediatric CRS (4701), Durham, North Carolina
  - The Children's Hospital of Philadelphia IMPAACT CRS (6701), Philadelphia, Pennsylvania
  - St. Jude/UTHSC CRS (6501), Memphis, Tennessee
  - Texas Children's Hosp. CRS (3801), Houston, Texas
  - Harborview Medical Center NICHD CRS (5027), Seattle, Washington
  - Seattle Children's Hospital CRS (5017), Seattle, Washington
  - University of Washington NICHD CRS (5029), Seattle, Washington
- Puerto Rico (2):
  - San Juan City Hosp. PR NICHD CRS (5031), San Juan
  - University of Puerto Rico Pediatric HIV/AIDS Research (6601), San Juan

REFERENCES:
- [Background] Patel K, Hernan MA, Williams PL, Seeger JD, McIntosh K, Van Dyke RB, Seage GR 3rd; Pediatric AIDS Clinical Trials Group 219/219C Study Team. Long-term effectiveness of highly active antiretroviral therapy on the survival of children and adolescents with HIV infection: a 10-year follow-up study. Clin Infect Dis. 2008 Feb 15;46(4):507-15. doi: 10.1086/526524. PMID 18199042
- [Background] Brady MT, Oleske JM, Williams PL, Elgie C, Mofenson LM, Dankner WM, Van Dyke RB; Pediatric AIDS Clinical Trials Group219/219C Team. Declines in mortality rates and changes in causes of death in HIV-1-infected children during the HAART era. J Acquir Immune Defic Syndr. 2010 Jan;53(1):86-94. doi: 10.1097/QAI.0b013e3181b9869f. PMID 20035164